CLINICAL TRIAL: NCT04206852
Title: Safety and Efficacy of Balloon Pulmonary Angioplasty in China
Status: Recruiting | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: BPA registry
Record Dates: First submitted 2019-10-26; First posted 2019-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Balloon pulmonary angioplasty — Balloon pulmonary angioplasty is an interventional technique where a balloon catheter is used to recanalize affected segments of pulmonary arteries identified during angiography.
  Other Names: BPA

SUMMARY:
Balloon pulmonary angioplasty (BPA) is a potential treatment for non-operable patients with chronic thromboembolic pulmonary hypertension (CTEPH).

The aim of this study was to evaluate the safety and efficacy of BPA in CTEPH patients not amenable to pulmonary endarterectomy(PEA) or suffered from persistent CTEPH after PEA.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, long-term observational project to study the safety and efficacy of BPA. Clinical evaluation, including: functional capacity, 6-minutes walking test, biomarkers, cardiopulmonary exercise test, electrocardiography, echocardiography, haemodynamics, pulmonary angiography and lung scintigraphy was performed before the initiation therapy of BPA, and 3-12 months after last session of BPA.

we also aim to evaluate the value of FAPI in predicting the efficacy and the prognosis of patients with CTEPH who received BPA.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with CTEPH according to ESC Guidelines (1) Mean PAP ≥ 25mmHg at rest; or if mean PAP < 25mmHg at rest, have exercise limitations from chronic thromboembolic disease (2)Abnormal ventilation perfusion lung scanning (VQ) scan, pulmonary angiogram, computer tomographic pulmonary angiogram, or magnetic resonance pulmonary angiogram confirming chronic thromboembolic disease as recommended by standard guidelines
2. Treatment with anticoagulation for ≥ 3 months before diagnosis of CTEPH
3. Not amenable to pulmonary endarterectomy
4. Willing to provide informed consent

Exclusion Criteria:

1. Patients unwilling or unable to provide written consent for participation in the study.
2. Impossible to follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic thromboembolic pulmonary hypertension patients admitted in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2028-05-11 (Estimated); Study Completion 2028-05-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of BPA procedure. | From initiation of BPA to 3-12 months after last session
  Surveillance of complications including: vessel injury, desaturation, cough, mild hemoptysis (<50ml), severe hemoptysis (>50ml), reperfusion pulmonary injury, death.
Change of Pulmonary artery pressure in mmHg caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  Pulmonary artery pressure in mmHg is obtained by right cardiac catheterization.
Change of Pulmonary vascular resistance (PVR) in Wood U caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  Pulmonary vascular resistance (PVR) in Wood U is obtained by right cardiac catheterization.
Change of cardiac index (CI) in L/m^2 caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  Cardiac index (CI) in L/m^2 is obtained by right cardiac catheterization.
Change of World Health Organization (WHO) functional capacity classification caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  World Health Organization is obtained from electronic medical records.
Change of six minutes walk distance in meter caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  World Health Organization is obtained from electronic medical records.
Change of N-terminal B-type natriuretic peptide in pg/ml caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  World Health Organization is obtained from electronic medical records.
Change of Peak VO2/kg in ml/min/kg caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  Peak VO2/kg in ml/min/kg is obtained by cardiopulmonary exercise test.
Change of diffusing capacity for carbon monoxide caused by series of BPA. | From initiation of BPA to 3-12 months after last session
  diffusing capacity for carbon monoxide in % is obtained from pulmonary function test
Change of fibroblast activation protein inhibitor expression after BPA | From initiation of BPA to 3-12 months after last session
  Change of fibroblast activation protein inhibitor expression after BPA

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - center of pulmonary vascular disease, Fuwai hospital, Beijing
  - Chinese Academy of Medical Sciences Fuwai hospital, Beijing